CLINICAL TRIAL: NCT05843864
Title: Utilizing Photobiomodulation Therapy for the Treatment of Lower Extremity Stress Fractures in a Military Training Setting
Brief Title: Photobiomodulation Therapy for the Treatment of Lower Extremity Stress Fractures in a Military Training Setting
Acronym: PM12
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Collaborators: The Geneva Foundation (Other); Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dan Rhon, Director, Musculoskeletal Research in Primary Care Program, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C.2023.025
Record Dates: First submitted 2023-04-18; First posted 2023-05-06 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Metatarsal Stress Fracture; Stress Fracture of Tibia
Keywords: Lower Extremity Bone Stress Injuries; Photobiomodulation; Military Populations; Photomedicine; Bone Stress Injuries
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard Physical Therapy and Photobiomodulation Therapy (Experimental): 61 Participants will be randomized to this group and will receive Photobiomodulation Therapy (PBMT) in addition to standard physical therapy.
  Interventions: Device: Photobiomodulation Therapy with Standard Physical Therapy
- Standard Physical Therapy and Sham Photobiomodulation Therapy (Sham Comparator): 61 Participants will be randomized to this group and will receive sham Photobiomodulation Therapy (PBMT) in addition to standard physical therapy.
  Interventions: Other: Sham Photobiomodulation Therapy with Standard Physical Therapy

INTERVENTIONS:
Device: Photobiomodulation Therapy with Standard Physical Therapy — Photobiomodulation Therapy (PBMT) will be provided by a trained individual in addition to standard physical therapy. Treatment will be delivered for approximately 10-16 minutes. Participants will then be instructed to rest for 5 minutes after the treatment.
  Other Names: Omnilux Plus 830
  Arms: Standard Physical Therapy and Photobiomodulation Therapy
Other: Sham Photobiomodulation Therapy with Standard Physical Therapy — Sham Photobiomodulation Therapy (PBMT) will be provided by a trained to the some location and with the same contact time and frequency as the active intervention (PBMT) in addition to standard physical therapy. Participants will then be instructed to rest for 5 minutes after the treatment.
  Arms: Standard Physical Therapy and Sham Photobiomodulation Therapy

SUMMARY:
The goal of this clinical trial is to compare photobiomodulation therapy (PBMT) in addition to standard of care in the treatment of tibial and metatarsal bone stress injuries in a military training setting.

Participants will all receive usual care and also be randomized to either active or sham photobiomodulation therapy. Effectiveness will be assessed based on time to return to duty and measures of pain and function.

* Participants will receive care for a maximum of 6 weeks.
* Participants will have follow-up through 4 months (or graduation/dismissal from training, whichever comes first).

DETAILED DESCRIPTION:
Trainees with a diagnosis of medial tibial or metatarsal bone stress injuries/stress fracture will be recruited. Patients that consent and enroll will be randomized to receive standard of care physical therapy with (1) photobiomodulation therapy (PBMT) or (2) sham PBMT. Patients will receive treatment 3x per week for up to 6 weeks. The primary outcome will be the time to return to duty. Secondary outcomes will include additional time points (3-week, 6-week, 4-month) and Patient-Reported Outcomes Measurement Information System (PROMIS®) measures of pain and function, lower extremity imaging and various other measures outlined in the "Outcome Measure" section. Participants will be asked to report any mineral supplementation and to record daily activity in a log. Survival analysis will be used to evaluate return to duty between treatment arms with censoring beyond 4 months.

Longitudinal hierarchical/multilevel models with random effects will be used to evaluate differences between treatment arms for the relevant outcome measures. Sensitivity analyses will be conducted predicting change in measures at the final follow-up relative to baseline, and will use linear generalized additive models.

ELIGIBILITY:
Inclusion Criteria:

* between ages 17-64 (inclusive) years old
* Currently completing Advanced Individual Training (AIT) training at Fort Sam Houston and at least 6 weeks prior to graduation
* Clinical diagnosis of metatarsal or medial tibial bone stress injury/stress fracture (unilateral or bilateral) by a healthcare provider based on accepted diagnostic criteria, with diagnostic imaging confirmation
* Able to read and understand English language for consent purposes
* Able to commit to study intervention and follow-up

Exclusion Criteria:

* Stress fracture to tibia that is not medial (e.g., anterior) or any location other than 5th metatarsal or medial tibia
* Has already become a severe non-union bone stress injury/fracture
* Received dry needling within the past 4 weeks
* Received Platelet Rich Plasma (PRP) injection, corticosteroid injection, or prolotherapy within the past 3 months
* Diagnosis of neuropathy affecting sensation to pain
* Current or chronic sciatica (lumbosacral radiculopathy) resulting in chronic or intermittent lower extremity pain, numbness, or tingling (all below the knee)
* Current or previous diagnosis of eating disorder (e.g., bulimia nervosa, anorexia nervosa, disordered eating, or other eating disorder not specified)
* Diagnosis of porphyria (light induced allergy) or photosensitive eczema
* Diagnosis of autoimmune disease (e.g., Lupus)
* Albinism
* Current use of anti-inflammatory steroids due to increased risk of Bone Stress Injury (BSI) with the past two weeks
* Current use of medications associated with sensitivity to heat or light in the past five days (e.g., amiodarone, chlorpromazine, doxycycline, hydrochlorothiazide, nalidixic acid, naproxen, piroxicam, tetracycline, thioridazine, voriconazole)
* Previous or current (within the past 2 years) use of Depo Provera
* Current use of pacemaker
* Tattoo in the area of treatment due to sensitivity to Photobiomodulation Therapy (PBMT)
* Concurrent participation in another research study receiving treatment for metatarsal or medial tibial bone stress injury/stress fracture
* Currently pregnant or plan to become pregnant during intervention period (safety of PBMT not established in pregnancy)
* Current diagnosis or symptoms of amenorrhea (≥ 6 months without a menstrual period) or oligomenorrhea (only 4-9 menstrual periods in a year)

Ages: 17 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 105 (Actual)
Dates: Start 2023-06-07 (Actual); Primary Completion 2025-03-25 (Actual); Study Completion 2025-08-14 (Actual)

PRIMARY OUTCOMES:
Time to Return to Duty | 4 months
  After treatment for stress fracture begins, the number of days before they return to duty will be counted.

SECONDARY OUTCOMES:
Defense and Veteran's Pain Rating Scale (DVPRS) with supplemental questions | Weekly up to 6 weeks, 4 months
  Pain will be captured weekly with this single-item assessment that utilizes a numerical rating scale (0-10, with 0 being "No Pain" and 10 being "As bad as it could be, nothing else matter") enhanced by functional word descriptors, color coding, and pictorial facial expressions matched to pain levels.
Percussion Test | Baseline
  The tester uses 2-3 fingers to firmly tap up and down on the injury area 3-4 times. Immediately afterwards, the individual provides a pain rating (Defense and Veterans Pain Rating Scale 0-10, with 0 being "No Pain" and 10 being "As bad as it could be, nothing else matter").
Percussion Test | 3 weeks
  The tester uses 2-3 fingers to firmly tap up and down on the injury area 3-4 times. Immediately afterwards, the individual provides a pain rating (Defense and Veterans Pain Rating Scale 0-10, with 0 being "No Pain" and 10 being "As bad as it could be, nothing else matter").
Percussion Test | 6 weeks
  The tester uses 2-3 fingers to firmly tap up and down on the injury area 3-4 times. Immediately afterwards, the individual provides a pain rating (Defense and Veterans Pain Rating Scale 0-10, with 0 being "No Pain" and 10 being "As bad as it could be, nothing else matter").
Percussion Test | 4 months
  The tester uses 2-3 fingers to firmly tap up and down on the injury area 3-4 times. Immediately afterwards, the individual provides a pain rating (Defense and Veterans Pain Rating Scale 0-10, with 0 being "No Pain" and 10 being "As bad as it could be, nothing else matter").
Hopping Test | Baseline
  Participants will be asked to perform up to 10 hops as tolerated on their symptomatic leg(s). At the conclusion of the test, participants will be asked to provide a pain rating (Defense and Veterans Pain Rating Scale 0-10, with 0 being "No Pain" and 10 being "As bad as it could be, nothing else matter"). If they are unable to reach 10 hops due to pain that will be recorded as an "incomplete".
Hopping Test | 3 weeks
  Participants will be asked to perform up to 10 hops as tolerated on their symptomatic leg(s). At the conclusion of the test, participants will be asked to provide a pain rating (Defense and Veterans Pain Rating Scale 0-10, with 0 being "No Pain" and 10 being "As bad as it could be, nothing else matter"). If they are unable to reach 10 hops due to pain that will be recorded as an "incomplete"
Hopping Test | 6 weeks
  Participants will be asked to perform up to 10 hops as tolerated on their symptomatic leg(s). At the conclusion of the test, participants will be asked to provide a pain rating (Defense and Veterans Pain Rating Scale 0-10, with 0 being "No Pain" and 10 being "As bad as it could be, nothing else matter"). If they are unable to reach 10 hops due to pain that will be recorded as an "incomplete"
Hopping Test | 4 months
  Participants will be asked to perform up to 10 hops as tolerated on their symptomatic leg(s). At the conclusion of the test, participants will be asked to provide a pain rating (Defense and Veterans Pain Rating Scale 0-10, with 0 being "No Pain" and 10 being "As bad as it could be, nothing else matter"). If they are unable to reach 10 hops due to pain that will be recorded as an "incomplete"
Lower Extremity Functional Scale (LEFS) | Baseline
  The LEFS is a self-reported assessment of physical function. It asks 20 questions with response options of "Extreme difficulty or unable to perform activity" (0), "Quite a bit of difficulty" (1), "Moderate difficulty" (2), "A little bit of difficulty" (3), "No difficulty" (4).
Lower Extremity Functional Scale (LEFS) | 3 weeks
  The LEFS is a self-reported assessment of physical function. It asks 20 questions with response options of "Extreme difficulty or unable to perform activity" (0), "Quite a bit of difficulty" (1), "Moderate difficulty" (2), "A little bit of difficulty" (3), "No difficulty" (4).
Lower Extremity Functional Scale (LEFS) | 6 weeks
  The LEFS is a self-reported assessment of physical function. It asks 20 questions with response options of "Extreme difficulty or unable to perform activity" (0), "Quite a bit of difficulty" (1), "Moderate difficulty" (2), "A little bit of difficulty" (3), "No difficulty" (4).
Lower Extremity Functional Scale (LEFS) | 4 months
  The LEFS is a self-reported assessment of physical function. It asks 20 questions with response options of "Extreme difficulty or unable to perform activity" (0), "Quite a bit of difficulty" (1), "Moderate difficulty" (2), "A little bit of difficulty" (3), "No difficulty" (4).

OTHER OUTCOMES:
Fredericson grading system | Baseline
  Severity of the stress fracture is assessed from Magnetic Resonance Imaging by a radiologist. Severity is classified as Grade "1", "2", "3", "4a" or "4b", with "Grade 1" being the least severe.
Fredericson grading system | 6 week
  Severity of the stress fracture is assessed from Magnetic Resonance Imaging by a radiologist. Severity is classified as Grade "1", "2", "3", "4a" or "4b", with "Grade 1" being the least severe.
Fredericson grading system | 4 months
  Severity of the stress fracture is assessed from Magnetic Resonance Imaging by a radiologist. Severity is classified as Grade "1", "2", "3", "4a" or "4b", with "Grade 1" being the least severe.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Rhon, DSc, PhD, Principal Investigator — Uniformed Services University of the Health Sciences
Locations (1):
- Brooke Army Medical Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wood AM, Hales R, Keenan A, Moss A, Chapman M, Davey T, Nelstrop A. Incidence and Time to Return to Training for Stress Fractures during Military Basic Training. J Sports Med (Hindawi Publ Corp). 2014;2014:282980. doi: 10.1155/2014/282980. Epub 2014 Jan 21. PMID 26464890
- [Background] Waterman BR, Gun B, Bader JO, Orr JD, Belmont PJ Jr. Epidemiology of Lower Extremity Stress Fractures in the United States Military. Mil Med. 2016 Oct;181(10):1308-1313. doi: 10.7205/MILMED-D-15-00571. PMID 27753569
- [Background] Reis JP, Trone DW, Macera CA, Rauh MJ. Factors associated with discharge during marine corps basic training. Mil Med. 2007 Sep;172(9):936-41. doi: 10.7205/milmed.172.9.936. PMID 17937356
- [Background] Molloy JM, Pendergrass TL, Lee IE, Chervak MC, Hauret KG, Rhon DI. Musculoskeletal Injuries and United States Army Readiness Part I: Overview of Injuries and their Strategic Impact. Mil Med. 2020 Sep 18;185(9-10):e1461-e1471. doi: 10.1093/milmed/usaa027. PMID 32175566
- [Background] Kardouni JR, McKinnon CJ, Taylor KM, Hughes JM. Timing of Stress Fractures in Soldiers During the First 6 Career Months: A Retrospective Cohort Study. J Athl Train. 2021 Dec;56(12):1278-1284. doi: 10.4085/1062-6050-0380.19. Epub 2021 May 11. PMID 33975344
- [Background] Wentz L, Liu PY, Haymes E, Ilich JZ. Females have a greater incidence of stress fractures than males in both military and athletic populations: a systemic review. Mil Med. 2011 Apr;176(4):420-30. doi: 10.7205/milmed-d-10-00322. PMID 21539165
- [Background] Lee D; Armed Forces Health Surveillance Center (AFHSC). Stress fractures, active component, U.S. Armed Forces, 2004-2010. MSMR. 2011 May;18(5):8-11. No abstract available. PMID 21793616

DOCUMENTS (1):
  • Informed Consent Form (2023-09-14): https://cdn.clinicaltrials.gov/large-docs/64/NCT05843864/ICF_000.pdf